CLINICAL TRIAL: NCT02893852
Title: Effects of the Cognitive Orientation to Daily Occupational Performance Approach on Activity and Participation of Brazilian Children With Developmental Coordination Disorder
Brief Title: Effects of CO-OP Approach on Activity and Participation of Brazilian Children With Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Clarice Ribeiro Soares Araujo, Doctoral Candidate, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE54543216.3.0000.5149/1.520
Record Dates: First submitted 2016-08-31; First posted 2016-09-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Motor Skills Disorders; Attention Deficit and Disruptive Behavior Disorders
MeSH Terms: conditions — Motor Skills Disorders; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- standard CO-OP Approach (Active Comparator): Task oriented and client-centred intervention with 12 sessions (10 interventional and 2 assessment sessions) with children and parents.
  Interventions: Behavioral: standard CO-OP Approach
- standard CO-OP Approach plus coaching parents (Experimental): Task oriented and client-centred intervention with 12 sessions (10 interventional and 2 assessment sessions) with children and parents with a "boost" of 4 group sessions of coaching for parents in groups.
  Interventions: Behavioral: standard CO-OP Approach plus coaching parents

INTERVENTIONS:
Behavioral: standard CO-OP Approach — The CO-OP protocol originally developed by Mandich and Polatajko (2004) comprises 12 sessions. The therapist teaches the participants a global cognitive strategy: GOAL - PLAN - DO - CHECK. The participants use the global strategy and cooperate to learn specific strategies to solve each task performance breakdown identified through Dynamic Performance Analyses (DPA). The therapist uses DPA at pre-intervention and throughout the sessions and mediational techniques to guide participants to use GOAL-PLAN-DO-CHECK to discover specific strategies to solve performance problems and to support generalization and transfer of skills.
  Other Names: CO-OP Approach
  Arms: standard CO-OP Approach
Behavioral: standard CO-OP Approach plus coaching parents — CO-OP Approach with parents coaching groups will include an addition of four extra coaching groups sessions for parents to provide additional information to supplement their knowledge on CO-OP (how to use GOAL-PLAN-DO-CHECK at home; how to use dynamic performance analysis to support their children's' performance solutions; to talk about their experiences with their children at home).
  Other Names: CO-OP Approach boosted
  Arms: standard CO-OP Approach plus coaching parents

SUMMARY:
The purpose of this study is to investigate the effects of the Cognitive Orientation to daily daily Occupational Performance Approach (CO-OP Approach) on activity and participation in school-aged children with developmental coordination disorder (DCD).

DETAILED DESCRIPTION:
Children with difficulty performing activities that reflect negatively on participation can meet the criteria for Developmental Coordination Disorder (DCD), which might impact their lives, leading to social isolation, depression and anxiety. Several studies have examined the effectiveness of different intervention approaches, including process-oriented approaches that focus on enhancing body functions and structures to improve performance on functional tasks. Although pediatric occupational therapists have traditionally used such approaches, evidence strongly suggests effectiveness for task-oriented interventions that focus on the performance of tasks that the child finds difficult to do. Among these, CO-OP Approach showed strong treatment effects. In CO-OP Approach, therapists use mediational techniques to teach cognitive strategies to improve occupational performance in goals chosen by the children. There is a need to examine systematic intervention alternatives for Brazilian children with DCD, and only one study examined occupational therapy intervention strategies for children with DCD.

The main purpose of the study is to examine the effects of two intervention models based on CO-OP Approach. The investigators will examine if a boosting on parent's engagement in CO-OP can improve skill acquisition, generalization and transfer in children with DCD. A pre-post design will be used and two groups will be included in this study (1) one receiving standard CO-OP Approach, (2) one receiving standard CO-OP Approach and an addition of coaching sessions in groups for parents. Follow-up data will be collected 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* score on MABC-2 below the 15th percentile;
* score on DCDQ-Brazil below age expectation, indicating problems on everyday living and/or academic skills;
* cognitive development within the expected age range according to the Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV);
* no diagnosis or signs of neurological or neuromuscular diseases.

Exclusion Criteria:

* no reading ability;
* child refuses to participate on assessment sessions.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-05-12; Primary Completion 2017-12-18 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Changes on the Canadian Occupational Performance Measure (COPM) | Changes on perceived performance and satisfaction from baseline to 12 weeks; Changes on perceived performance and satisfaction from baseline to 24 weeks, and changes on perceived performance from post intervention to 24 weeks.
Changes on frequency on the Participation and Environment Measure -Child and Youth (PEM-CY) | Changes on frequency levels of participation from baseline to 12 weeks; Changes on frequency levels of participation at baseline to 24 weeks, and changes on frequency levels of participation from post intervention to 24 weeks.
Changes on involvement on the Participation and Environment Measure -Child and Youth (PEM-CY) | Changes on involvement levels of participation from baseline to 12 weeks; Changes on involvement levels of participation from baseline to 24 weeks, and changes on involvement levels of participation from post intervention to 24 weeks.
Changes on the Performance Quality Rating Scale (PQRS) | Changes on actual performance from baseline to 12 weeks; Changes on actual performance from baseline to 24 weeks, and changes on actual performance from post intervention to 24 weeks.

SECONDARY OUTCOMES:
Changes on Motor Assessment Battery for Children Second Edition (MABC2) | Changes on motor proficiency from baseline to 12 weeks.
Changes on Five Digits Test (FDT) | Changes on Cognitive flexibility from baseline to 12 weeks.
Changes on the Self-Perception Profile for children | Changes on self-perception from baseline to 12 weeks; Changes on self-perception from baseline to 24 weeks, and changes on self-perception from post intervention to 24 weeks.
Changes on Tower of London Test (TOL) | Changes on mental planning from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Livia C Magalhaes, PhD, Study Chair — Federal Unversity of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Thornton A, Licari M, Reid S, Armstrong J, Fallows R, Elliott C. Cognitive Orientation to (Daily) Occupational Performance intervention leads to improvements in impairments, activity and participation in children with Developmental Coordination Disorder. Disabil Rehabil. 2016;38(10):979-86. doi: 10.3109/09638288.2015.1070298. Epub 2015 Jul 27. PMID 26213242
- [Background] Miller LT, Polatajko HJ, Missiuna C, Mandich AD, Macnab JJ. A pilot trial of a cognitive treatment for children with developmental coordination disorder. Hum Mov Sci. 2001 Mar;20(1-2):183-210. doi: 10.1016/s0167-9457(01)00034-3. PMID 11471396
- [Background] Missiuna C, Mandich AD, Polatajko HJ, Malloy-Miller T. Cognitive orientation to daily occupational performance (CO-OP): part I--theoretical foundations. Phys Occup Ther Pediatr. 2001;20(2-3):69-81. PMID 11345513
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506
- [Background] Levac D, Wishart L, Missiuna C, Wright V. The application of motor learning strategies within functionally based interventions for children with neuromotor conditions. Pediatr Phys Ther. 2009 Winter;21(4):345-55. doi: 10.1097/PEP.0b013e3181beb09d. PMID 19923975
- [Background] Polatajko HJ, Mandich AD, Miller LT, Macnab JJ. Cognitive orientation to daily occupational performance (CO-OP): part II--the evidence. Phys Occup Ther Pediatr. 2001;20(2-3):83-106. PMID 11345514
- [Background] Capistran J, Martini R. Exploring inter-task transfer following a CO-OP approach with four children with DCD: A single subject multiple baseline design. Hum Mov Sci. 2016 Oct;49:277-90. doi: 10.1016/j.humov.2016.07.004. Epub 2016 Aug 12. PMID 27522644
- [Background] Mandich AD, Polatajko HJ, Rodger S. Rites of passage: understanding participation of children with developmental coordination disorder. Hum Mov Sci. 2003 Nov;22(4-5):583-95. doi: 10.1016/j.humov.2003.09.011. PMID 14624835
- [Derived] Araujo CRS, Cardoso AA, Magalhaes LC. Efficacy of CO-OP Approach With and Without Parental Coaching: RCT Study Protocol: Efficacite de l'approche CO-OP avec et sans coaching parental : protocole d'essai clinique randomise. Can J Occup Ther. 2021 Jun;88(2):182-194. doi: 10.1177/00084174211005889. Epub 2021 Apr 13. PMID 33845626